CLINICAL TRIAL: NCT00517959
Title: Efficacy of Stereotactic Conformal Radiotherapy (SCRT) Compared to Conventional Radiotherapy in Minimising Late Sequelae in Children and Young Adults With Brain Tumours: a Randomised Clinical Trial
Brief Title: SCRT Versus Conventional RT in Children and Young Adults With Low Grade and Benign Brain Tumors
Acronym: SCRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Terry Fox Foundation (Other)
Responsible Party: Principal Investigator, Rakesh Jalali, Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRT Trial
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-06

CONDITIONS: Low Grade Gliomas; Craniopharyngioma; Ependymomas; Meningiomas
Keywords: Stereotactic radiotherapy; conformal radiotherapy; late sequelae; cognition; endocrine dysfunction
MeSH Terms: conditions — Craniopharyngioma; Ependymoma; Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Stereotactic conformal radiotherapy (SCRT)
  Interventions: Radiation: Stereotactic Conformal radiotherapy
- 2 (Other): Conventional radiotherapy Patients in this arm will be treated with conventional radiotherapy techniques being used at the moment in the department. This involves patient being immobilised with a customised thermoplastic mask after which they will have a contrast enhanced planning CT scan. The radiation oncologist will draw the tumour on the appropriate CT slices and a margin of 1-2 cms grown for the planning target volume. Beam arrangement will be relatively simple and typically consist of 2-3 coplanar fields using 6 MV photons. Conventional planning optimisation will be carried out by the use of wedges, beam weightage and corner shields as appropriate. Radiotherapy doses, prescription and fractionation schedules will be identical to the SCRT arm
  Interventions: Radiation: Conventional radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Conformal radiotherapy — SCRT
  Arms: 1
Radiation: Conventional radiotherapy
  Arms: 2

SUMMARY:
Brain tumours are the commonest solid tumours in children and the second most common neoplasms overall in this patient population. Radiotherapy plays an important part in the management in a majority of these tumours. While the cure rates of these tumours, especially the benign and low grade ones are quite encouraging, the treatment itself may lead to some late sequelae, which could have significant implications in the quality of life in these long-term survivors.

Stereotactic conformal radiotherapy (SCRT) is a modern high-precision radiotherapy technique, which reduces the volume of normal brain irradiated and has the capability to minimise the doses to critical structures. The present study is designed to prospectively estimate the incidence and severity of neuropsychological, cognitive and neuroendocrine dysfunction following radiotherapy delivered with conventional and stereotactic techniques and would be one of the most comprehensive studies providing very important longitudinal and reliable data regarding these sequelae. The study involving 200 patients would be to the best of our knowledge not only the largest ever study conducted so far but also the only randomised trial assessing these sequelae in patients receiving focal brain irradiation.

The study also examines whether the physical advantages of modern technological progress translate in clinical benefit. This could have significant implications in the radiotherapeutic management of children and young adults with brain tumours. The study is unique in design in terms of evaluating the efficacy of SCRT with respect to conventional radiotherapy in terms of long term tumour control and treatment related complications.

DETAILED DESCRIPTION:
1.0 BACKGROUND AND RATIONALE

Brain tumours are the commonest solid tumours in children and with appropriate treatment, nearly half of them achieve long term cure. Radiotherapy is essential in the management of a majority of these tumours. Conventional radiotherapy alone or in combination with surgery and/or chemotherapy in tumours such as optic gliomas, hypothalamic gliomas, craniopharyngiomas, germ cell tumours, and other low grade tumours achieves excellent long term control rates ranging from 70 to 95%. However, while the tumour control has been effective, there have been concerns about treatment related morbidity.

which included cognitive dysfunction in 38%, motor deficit in 25%, visual impairment in 20%, hormonal dysfunction in 20% and psychological-emotional problems in 14% of the survivors.

It is difficult to ascertain from these reports the exact contribution of each of these factors and how they interact with each other. Radiotherapy is believed to be at least partly responsible although its exact role is yet to be quantified. Most of the evidence regarding post-radiotherapy neuropsychological and cognitive dysfunction is from retrospective studies involving whole brain radiotherapy.

Neuroendocrine dysfunction is well-documented late sequelae following treatment of patients with brain tumours. This could either be due to direct involvement of the pituitary hypothalamic axis (PHA) by the tumour or as a result of surgical or radiation injury to this region. For tumours not directly involving the PHA, the commonest cause of neuroendocrine dysfunction is cranial irradiation. PHA region unavoidably receives radiation with whole brain radiotherapy or if the tumour itself is arising from this region. For the treatment of tumours adjacent to PHA but not involving it, it may be frequently a part of radiotherapy planning target volume, which includes the gross tumour and a margin to account for any microscopic disease and possible daily set up inaccuracies and thus receive significant doses. The region may also sometimes come in the entry / exit path of radiation beams during treatment of tumours even away from this region. Radiation induced hormonal abnormalities are generally dose dependent and may develop many years after irradiation. To reduce the impact of endocrine dysfunctions on physical, mental and sexual development, it is important to detect and treat them timely. Early growth hormone replacement is the only way to minimise growth retardation caused by its deficiency but the treatment is expensive with significant financial implications, especially in our country. The annual cost of GH replacement is approximately Rs 200,000.00, which is prohibitive for the vast majority of the Indian parents as is the cost of LHRH analogues, which is useful to prevent early epiphyseal fusion and stunted growth in children with post radiation or tumour related precocious puberty.

1.4 Evolution of Stereotactic conformal radiotherapy (SCRT) Conventional radiotherapy techniques generally involve the use of 2-3 radiation beams covering the tumour and a margin of 1-3 cms for any subclinical disease and physical inaccuracies in the daily treatment delivery. The last decade has seen tremendous technological advances in radiotherapy planning and accurate treatment delivery. Stereotactic radiosurgery (SRS) and stereotactic radiotherapy (SRT) techniques involve firm and accurate immobilisation with fixed or relocatable frames, high precision three-dimensional (3-D) target localisation with CT/CT-MRI fusion and focused radiation delivery. This is achieved either with a multiple source cobalt unit (gamma knife) or with multiple arcs using a modified conventional linear accelerator. Such conventional stereotactic irradiation techniques typically produce spherical high dose volumes and are therefore suitable only for small spherical lesions. A majority of the brain tumours considered for radiotherapy however are not spherical and frequently extend to adjacent structures. To treat large non-spherical volumes with conventional SRS requires the addition of multiple small spherical high dose volumes described as multiple isocentre treatment. The overlap of high dose spheres results in dose inhomogeneity, which has been associated with a higher incidence of radiation induced complications. It has been previously demonstrated that the optimum way of delivering high precision localised irradiation to larger non-spherical targets is with the use of multiple conformal fixed fields with individualised shielding of each radiation field conforming to the shape of the target. This principle of conformal therapy combined with the precision of stereotactic localisation and focused radiation delivery is described as stereotactic conformal radiotherapy (SCRT).

Traditionally, stereotactic irradiation has been delivered in a one session as single fraction radiosurgery. High doses of radiation given in one fraction are known to be associated with a high risk of radiation induced damage to normal tissue and this is particularly true for the central nervous system. Giving radiation in small individual doses allows the delivery of higher radiation doses without serious injury to the normal tissues, which is especially important for normal CNS structures. Single fraction SRS has been shown to be associated with considerable neurological toxicity to the optic apparatus the cranial nerves and normal brain. With the application of high precision relocatable non-invasive means of immobilisation, it has become possible to deliver stereotactic irradiation in a fractionated manner. The technique of SCRT combines the precision of focused radiation delivery and the radiobiological advantages of fractionation. It also ensures homogenous dose distribution within the irradiated volume further reducing the risk of damage.

The basic aim of high precision SCRT is to achieve a high dose differential between the tumour and the surrounding normal tissues. This allows for either an increase in the tumour dose to improve local control or for a potential decrease in radiation damage to the normal tissues. Further optimisation of the technique involving 3-4 conformal non-coplanar field arrangement has shown a significant dose reduction to the normal brain. Preliminary experience, mainly in adults has shown this technique to be feasible during the routine practice of a busy radiotherapy department. Early results in terms of local control are same as that with conventional radiotherapy, with an increased sparing of the surrounding normal brain and adjacent critical structures. While the experience is limited in young children, a few reports have suggested it to be feasible in this population also. The technique has the potential to minimise the dose to any critical site close to the tumour like pituitary-hypothalamic complex, cochlea, brain stem, optic apparatus and the mesial temporal lobes, which are believed to be the common sites of radiation injury leading to late morbidity.

NEED FOR THE PRESENT STUDY The finding of significant long-term effects in a large proportion of brain tumour survivors mandates the development of treatment strategies designed to minimise their impact on the quality of life. Although the precise role of radiotherapy in the causation of various post treatment sequelae is not established, it is generally believed to be at least partly responsible for these effects. There have been attempts to modify the management in terms of avoiding, delaying radiotherapy or reducing the total radiation dose to the tumour with a view to reduce its impact on the long-term toxicity. However, reduction of radiotherapy doses to the tumour has been shown to result in poorer local control rates. Also, a majority of the patients in whom the radiation is delayed eventually do require radiotherapy at later stages (37). There is also evidence that radiotherapy given upfront yields superior disease control than radiotherapy given at the time of tumour progression (38,39). In light of this data, there is therefore, an ever-increasing need to explore techniques of radiotherapy minimising the irradiation to the normal brain and critical structures without compromising radiotherapy doses essential for tumour control. SCRT is a modern high-precision radiotherapy technique, which reduces the volume of normal brain irradiated and has the capability to minimise the doses to critical structures.

The evidence of long term effects of focal irradiation so far is from retrospective studies and a few small prospective trials. There is therefore, a great need to evaluate this issue in a prospective manner in a large number of patients. The present study is designed to prospectively estimate the incidence and severity of neuropsychological, cognitive and neuroendocrine dysfunction following radiotherapy delivered with conventional and stereotactic techniques and would be one of the most comprehensive studies providing very important longitudinal and reliable data regarding these sequelae. The study involving 200 patients would be to the best of our knowledge not only the largest ever study conducted so far but also the only randomised trial assessing these sequelae in patients receiving focal brain irradiation.

The study also examines whether the physical advantages of modern technological progress translate in clinical benefit. This could have significant implications in the radiotherapeutic management of children and young adults with brain tumours. The study is unique in design in terms of evaluating the efficacy of SCRT with respect to conventional radiotherapy in terms of long term tumour control and treatment related complications.

If the present trial succeeds in reducing the incidence and severity of radiotherapy related sequelae by SCRT technique, it would undoubtedly result in a tremendous benefit to these patients. A possible reduction in the neuroendocrine sequelae not only will improve the quality of life of the patients but would also result in major financial saving. This is critical in patients living in the developing countries where the cost of endocrinological management in terms of hormonal assays and their replacement is largely prohibitive.

We have until Januray 2009 accrued 128 patients so far in the trial

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary intracranial tumours such as low-grade glioma, meningioma, craniopharyngiomas, ependymomas and other benign tumours considered for radical focal radiotherapy.
2. Tumours measuring upto 7 cms on maximum dimension on the CT/MRI.
3. Age 3 to 25 years.
4. NPS of 0-3.
5. Informed consent from patients or parents as appropriate.
6. Long-term follow up expected

Exclusion Criteria:

1. Previous radiotherapy.
2. Planned adjuvant chemotherapy.
3. Expected median survival of less than two years.
4. Patient not cooperative for planning and execution of SCRT.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2001-05; Primary Completion 2013-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of neuropsychological and neuroendocrine function in the two arms

SECONDARY OUTCOMES:
Progression free and overall survival. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Jalali, MD, Principal Investigator — Tata Memorial Hospital; Rajiv Sarin, MD FRCR, Principal Investigator — ACTREC, TMC
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

REFERENCES:
- [Result] Jalali, Goswami S, Sarin R, More N, Siddha M and Kamble R . Int J of Radiat Oncol Biol Physics 2006;66(4):S14-S19.
- [Derived] Jalali R, Ghosh S, Chatterjee A, Goswami S, Shah N, Dutta D, Krishna U, Gupta T, Goda JS. High-precision radiotherapy achieves excellent long-term control and preserves function in pediatric craniopharyngioma-Subset analysis of a randomized trial. Neuro Oncol. 2025 Sep 17;27(8):2147-2157. doi: 10.1093/neuonc/noaf049. PMID 40056158
- [Derived] Chatterjee A, Goda JS, Gupta T, Kamble R, Mokal S, Krishnatry R, Sarin R, Jalali R. A randomized trial of stereotactic versus conventional radiotherapy in young patients with low-grade brain tumors: occupational therapy-based neurocognitive data. Neurooncol Adv. 2020 Oct 1;2(1):vdaa130. doi: 10.1093/noajnl/vdaa130. eCollection 2020 Jan-Dec. PMID 33235996
- [Derived] Jalali R, Gupta T, Goda JS, Goswami S, Shah N, Dutta D, Krishna U, Deodhar J, Menon P, Kannan S, Sarin R. Efficacy of Stereotactic Conformal Radiotherapy vs Conventional Radiotherapy on Benign and Low-Grade Brain Tumors: A Randomized Clinical Trial. JAMA Oncol. 2017 Oct 1;3(10):1368-1376. doi: 10.1001/jamaoncol.2017.0997. PMID 28570730